CLINICAL TRIAL: NCT05333003
Title: Semaglutide in Comorbid Schizophrenia Spectrum Disorder and Obesity for Metformin Non-responders: a Single-blind Randomized Control Trial
Brief Title: Semaglutide in Comorbid Schizophrenia Spectrum Disorder and Obesity
Acronym: Sema
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Margaret Hahn, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 139/2020
Record Dates: First submitted 2022-03-25; First posted 2022-04-18 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Schizophrenia Spectrum Disorders
Keywords: Schizophrenia spectrum disorders; GLP-1 receptor agonists; Weight; Antipsychotics
MeSH Terms: conditions — Body Weight | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide (Experimental): Semaglutide medication will be taken by participants on a weekly schedule, and adherence tracked
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): Placebo will be taken by participants on a weekly schedule, and adherence tracked
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Semaglutide — The semaglutide dose will start with 0.25 mg/week, and slowly increased every four weeks as tolerated up to a maximal dose of 2 mg/week
  Arms: Semaglutide
Other: Placebo — Placebo will be provided to participants
  Arms: Placebo

SUMMARY:
Rates of obesity in patients with schizophrenia-spectrum disorder (SSD)s have reached epidemic proportions, with established contributing effects of antipsychotic (AP) medications. Among agents approved for chronic weight management, glucagon-like peptide-1 receptor agonists (GLP-1RA) are associated with reductions in cardiovascular mortality, with recent FDA approval for once weekly semaglutide for this indication. This study will investigate whether semaglutide is effective in reducing body weight in overweight or obese individuals with SSDs who are on APs and do not demonstrate adequate weight loss on metformin (the first line treatment for weight loss in SSDs).

DETAILED DESCRIPTION:
People with SSDs die early of iatrogenic cardiometabolic disease. Clinically, metformin remains the first line agent to mitigate this risk. In real-world clinical practice, metformin is likely to remain the first line treatment for AP-induced weight gain (given low cost, efficacy, and safety data). However, metformin is only effective in ~20% of patients. Hence, there is a need for interventions for AP-induced weight gain non-responsive to metformin. GLP-1RAs might represent the next rational step as they have a good safety profile, advantages of weekly administration, and early efficacy evidence to support their use in SSD and comorbid obesity, with benefits on dysglycemia, and visceral adiposity. Semaglutide, recently approved for chronic weight loss is an attractive option given a similar adverse effect profile but superior metabolic efficacy compared to other GLP-1 agents. The observations supporting an association between metabolic perturbations and cognition, along with preliminary evidence for neuroprotective effects of GLP-1RAs, suggest that by modifying metabolic risk factors, the investigators may be able to target difficult-to-treat domains of the illness such as cognitive dysfunction.

This study will examine the effect of semaglutide on:

1. Percentage change in body weight
2. Measures of glucose metabolism and cardiovascular risk factors
3. Psychopathology
4. Cognition
5. Lifestyle-based assessments

ELIGIBILITY:
Inclusion Criteria:

* Stable outpatients or inpatients aged 18-70 years, diagnosed with schizophrenia spectrum disorder, or major depressive disorder with psychotic features, or bipolar disorder (does not need to have psychotic features)
* On maintenance treatment with an AP (stable dose for ≥3 months)
* BMI must be ≥30 kg/m2, OR ≥27 kg/m2 with the presence of at least one weight-related comorbidity (treated or untreated): hypertension, dyslipidaemia, obstructive sleep apnea, or impaired fasting glucose, OR BMI ≥25 with individual having gained >5% bodyweight in association with AP treatment
* History of either failure to tolerate metformin or failure to lose ≥5% body weight over at least 16 weeks on the highest tolerated trial of metformin, and who are not currently being treated with metformin (minimum of 1 week metformin-free prior to study entry)

Exclusion Criteria:

* Patients with severe substance disorder other than tobacco or caffeine use disorder; only severe substance use disorder is exclusionary for cannabis use
* Liver, or renal dysfunction
* A positive drug urine screen other than cannabis as per PI discretion
* Sexually active females of child-bearing age not on a regular contraceptive, or nursing or with a positive pregnancy test
* Clinical or laboratory evidence of uncompensated cardiovascular, endocrine, haematological, or pulmonary disease
* History of reactive hypoglycaemia
* Treatment within 3 months, or failure to tolerate GLP-1RA
* Type 1 Diabetes (T1D) or current diagnosis of Type 2 Diabetes (T2D), diagnosis of T2D on OGTT screen, or HbA1c > 6.5%
* Use of Health Canada approved weight-lowering agents, warfarin, coumarin derivatives, or medication with significant renal impact
* Major medical or surgical event within the preceding 3 months
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome
* History of pancreatitis or elevated amylase on screen
* History of severe gastrointestinal disease, (i.e. gastroparesis)
* Acute suicidal risk
* Uncompensated thyroid disorder
* History of heart rhythm disturbances, conduction system abnormalities, or evidence of clinically relevant abnormalities on screening ECG.
* Any condition that interferes with the safe acquisition of MRI data such as metal implants, pacemakers, aneurysm clips, cochlear implants (only for the MRI component; can participate in the remainder of the trial)
* History of gallstones with intact gallbladder or those at increased risk of gallbladder complications (with intact gallbladder)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Weight change | 32 weeks
  Percentage change in body weight (kg)

SECONDARY OUTCOMES:
Body Mass Index (BMI) | 32 weeks
  A person's weight in kilograms divided by height in metres squared
Waist circumference | 32 weeks
  Measured in centimetres
Oral glucose tolerance test | 32 weeks
  A standard glucose drink (75g) is given orally, and bloodwork containing insulin (pmol/L) and glucose (mmol/L) levels are obtained both at baseline and 2 hours after the glucose drink. These measures will help indicate B cell function and whole body insulin sensitivity, allowing for the proportion of individuals converting to impaired glucose tolerance, prediabetes, or type 2 diabetes to be determined.
Visceral and hepatic adiposity | 32 weeks
  An abdominal surface coil on the MRI will be used for this body composition measure
Fasting lipid profile | 32 weeks
  Cholesterol, high-density lipoprotein (HDL), low-density lipoprotein (LDL) and triglyceride levels will be collected through bloodwork in mmol/L
Psychopathology - Brief Psychiatric Rating Scale (BPRS) | 32 weeks
  Structured scale used to measure psychiatric symptoms
Psychopathology - Calgary Depression Scale for Schizophrenia (CDSS) | 32 weeks
  Structured scale used to measure depression in schizophrenia
Psychopathology - Global Assessment of Functioning (GAF) | 32 weeks
  Structured scale used to rate the global functioning of patient
Psychopathology - Clinical Global Impression scale (CGI) | 32 weeks
  Structured scale used to rate the global impression of patient
Change in cognitive performance | 32 weeks
  Evaluated through a standard scale called the MATRICS Consensus Cognitive Battery (MCCB)
Lifestyle assessment - Assessment of Quality of life (AQoL) | 32 weeks
  A structured scale used to measure health-related quality of life
Lifestyle assessment - WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) | 32 weeks
  A structured measure of health and disability
Lifestyle assessment - International Physical Activity Questionnaire (IPAQ) | 32 weeks
  A structured measure of physical activity practices
Lifestyle assessment - The Fagerstrom Test of Nicotine Dependence (FTND) | 32 weeks
  A structured scale used to measure the intensity of nicotine dependence related to cigarette smoking
Lifestyle assessment - Penn State Nicotine Dependence Index-Cigarette/Electronic Cigarette | 32 weeks
  A structured measure used to quantify the intensity of physical dependence across various nicotine products
Lifestyle assessment - Canadian Diet History Questionnaire II (C-DHQ II) | 32 weeks
  A structured, comprehensive questionnaire used to measure food frequency
Lifestyle assessment - Food Cravings Questionnaire (FCQ) | 32 weeks
  A structured item used to measure frequency and intensity of food cravings

OTHER OUTCOMES:
Structural MRI | 32 weeks
  High-resolution anatomical image of the brain will be acquired
Resting state functional MRI (rsfMRI) | 32 weeks
  The resting-state echo-planar imaging will be used to analyze fronto-temporal network connectivity
Arterial spin labeling (ASL) | 32 weeks
  This scan will be performed to assess the effects on cerebral blood flow
1H-Magnetic resonance spectroscopy (MRS) | 32 weeks
  A single voxel spectra will be acquired for a volume of interest placed over the bilateral striatum, to measure glutamate levels

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Hahn, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada